CLINICAL TRIAL: NCT07016854
Title: Evaluation of Early Endovascular Treatment in Acute Ischemic Stroke With Isolated Internal Carotid Artery Occlusion (EVT-iICAO)
Brief Title: Early Endovascular Treatment in Isolated Internal Carotid Artery Occlusion
Acronym: EVT-iICAO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EVT-iICAO
Record Dates: First submitted 2025-05-25; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Stroke, Acute Ischemic
Keywords: endovascular treatment; isolated internal carotid artery occlusion
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endovascular treatment plus the best medical treatment (Experimental)
  Interventions: Procedure: Endovascular treatment; Drug: The best medical treatment
- The best medical treatment (Active Comparator)
  Interventions: Drug: The best medical treatment

INTERVENTIONS:
Procedure: Endovascular treatment — Endovascular treatment could be performed with any recanalization strategy, such as thrombectomy with aspiration or stent and angioplasty with balloon dilation or stent implantation, depending on the operator's choice and anatomical and radiological circumstances. In the setting of emergency stenting, the use of antiplatelet agents will depend on operator preference, anatomy, and bleeding risk.
  Arms: Endovascular treatment plus the best medical treatment
Drug: The best medical treatment — Medical treatment includes intravenous thrombolysis, anticoagulant or antiplatelet drugs, etc. which is determined by the attending physician according to the Chinese guidelines or expert consensus.

SUMMARY:
The primary hypothesis being tested in this trial is that acute ischemic stroke with isolated internal carotid artery occlusion will have improved clinical outcomes when given early endovascular treatment compared with that of given best medical treatment.

DETAILED DESCRIPTION:
Stroke is the leading cause of death and disability among Chinese residents, and ischemic stroke accounts for 70-80% of all strokes. Isolated internal carotid artery occlusion (iICAO) refers to occlusion of the internal carotid artery, which is not involve the circle of Willis, the M1 and the proximal M2 segment of the middle cerebral artery. IICAO accounts for about 20-25% of symptomatic acute internal carotid artery occlusion. Previous studies have shown that despite the best medical treatment, including intravenous thrombolysis, the early recanalization rate of patients with acute iICAO is only 4.4%-23%, and less than half of the patients eventually achieve self-care. Endovascular Treatment (EVT) is the most effective reperfusion therapy for large vessel occlusive stroke. Since only a few retrospective studies have reported the efficacy and safety of early EVT in patients with acute iICAO stroke, there is a lack of high-level prospective evidence so far. Therefore, the aim of this study is to conduct a prospective, multicenter, open-label, randomized controlled clinical trial to evaluate the efficacy and safety of early EVT in patients with acute iICAO stroke.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18.
2. Clinical signs consistent with an acute ischemic stroke and randomization no later than 23 hours after the time last known to be well.
3. CTP, CTA or enhanced MRA within 1 hour before randomization showed that the offending vessel was isolated internal carotid artery occlusion, namely occlusion of C1-C6 segments (according to Bouthillier's segmentation) at any location. There was no ipsilateral intracranial branch occlusion (T or L shape of internal carotid artery, M1 or M2 segment of middle cerebral artery, A1 or A2 segment of anterior cerebral artery, P1 or P2 segment of posterior cerebral artery).
4. Neurological deficit with a NIHSS of >5, or ≤5 points with disabling symptoms (complete hemianopsia, severe aphasia, neglect, any limb weakness that cannot sustain resistance to gravity, and functional loss that is considered by doctors and patients to be potentially disabling by clinical evaluation).
5. Mismatch: target Mismatch Profile on CT perfusion or MRI (ischemic core volume is < 70 ml, mismatch ratio is ≥1.8 and mismatch volume is ≥15 ml); clinical-imaging mismatch defined as an ASPECTS score of more than 5, was present if perfusion data were not available or imaging quality was poor enough to be interpreted.
6. mRS Score before stroke ≤2.
7. Patient/Legally Authorized Representative has signed the Informed Consent form.

Exclusion Criteria:

1. The patient underwent carotid endarterectomy within 1 month.
2. Severe comorbid condition with life expectancy less than 6 months at baseline.
3. Other suspected cerebrovascular diseases (vasculitis, untreated cerebrovascular malformation, intracranial aneurysm, etc.) based on history and CTA/MRA.
4. Women who are pregnant or planning to become pregnant at the time of the study and who are known to be pregnant or breastfeeding at the time of admission.
5. Known life-threatening allergic reactions to contrast media or intravascular products.
6. Chronic internal carotid artery occlusion, defined as known carotid artery occlusion (imaging examination) ≥30 days before randomization or highly suspected chronic internal carotid artery occlusion based on medical history and CT/MRI.
7. Tandem occlusion, which was defined as internal carotid artery occlusion combined with large intracranial vessel occlusion (T or L shape of internal carotid artery, M1 or M2 segment of middle cerebral artery, A1 or A2 segment of anterior cerebral artery, P1 or P2 segment of posterior cerebral artery).
8. No known vascular access.
9. Suspected aortic dissection based on medical history, clinical evaluation or/and imaging.
10. Evidence of intracranial hemorrhage on CT/MRI.
11. Patient unable to come or unavailable for follow-up.
12. Pre-existing neurological or psychiatric disease that would confound the neurological or functional evaluations.
13. Seizures at stroke onset if they make the diagnosis of stroke doubtful and preclude obtaining an accurate baseline NIHSS assessment.
14. Patients have contraindications to the use of heparin and antiplatelet drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Good clinical outcome | 90（±14）days after randomization
  Score in modified Rankin Scale (mRS) ≤ 2

SECONDARY OUTCOMES:
National Institute of Health Score Scale (NIHSS) | 24（-6/+12）hours after randomization
Recanalization rate of internal carotid artery | 24（-6/+12）hours and 90（±14）days after randomization
Early neurologic improvement | 24 hours after randomization
  The NIHSS score of 0-2 at 24 hours or a decrease of ≥8 points from baseline
Early neurological deterioration | 24 hours or 5-7 days after randomization
  The NIHSS score at 24 hours or on 5-7 days increased by ≥4 points from baseline
Mortality | 90 days after randomization
  All-cause mortality
Symptomatic intracranial hemorrhage | 24（-6/+12）hours after randomization
Procedural/device-related adverse events | 30（±5）days after randomization

CONTACTS AND LOCATIONS:
Locations (1):
- Sir Run Run Shaw Hospital, Hangzhou, Zhejiang, China